CLINICAL TRIAL: NCT05005650
Title: Survival Impact of Internal Mammary or Supraclavicular Lymphadenectomy on Stage IVB Ovarian Cancer With Supradiaphragmatic Lymph Node Metastasis
Brief Title: Survival Impact of Internal Mammary or Supraclavicular Lymphadenectomy
Acronym: SDLNOC
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee Seung Kim, Associate Professor, Seoul National University Hospital
Other Study IDs: SDLNOC
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Cancer Stage IV; Lymph Node Metastases
Keywords: internal mammary lymph node; supraclavicular lymph node; cardiophrenic lymph node
MeSH Terms: conditions — Ovarian Neoplasms; Lymphatic Metastasis | interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: debulking surgery — debulking surgery as primary debulking surgery or interval debulking surgery

SUMMARY:
To evaluate the survival impact of extensive lymphadenectomy as part of debulking surgery in stage IVB ovarian cancer with supradiaphragmatic lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed ovarian, fallopian tubal, primary peritoneal cancer
* Patients suspected of metastatic lymph nodes in the cardiophrenic, internal mammary, and/or supraclavicular lymph node by CT (size larger than 5mm)
* Patients clinically diagnosed FIGO stage IVB ovarian, fallopian tubal, primary peritoneal cancer
* Patients underwent debulking surgery (primary debulking surgery or interval debulking surgery) at Seoul National University Hospital from January 2010 to January 2020
* Patients age 18-90

Exclusion Criteria:

* Borderline or benign ovarian disease
* Patient didn't undergo debulking surgery
* Non-epithelial ovarian cancer

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent treatment at University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From date of treatment until the date of first documented progression or date of death (by any cause, in the absence of disease progression) whichever came first, assessed up to 120 months
  the time interval from the treatment start date to disease recurrence or progression date

SECONDARY OUTCOMES:
Overall survival | From the date of treatment start date until death due to any cause, assessed up to 120 months
  the time interval from the treatment start date to death or end of study date

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Kim, Pf, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, 시/도/주, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Randall LM, Pothuri B. The genetic prediction of risk for gynecologic cancers. Gynecol Oncol. 2016 Apr;141(1):10-6. doi: 10.1016/j.ygyno.2016.03.007. PMID 27016223
- [Background] Ataseven B, Grimm C, Harter P, Heitz F, Traut A, Prader S, du Bois A. Prognostic impact of debulking surgery and residual tumor in patients with epithelial ovarian cancer FIGO stage IV. Gynecol Oncol. 2016 Feb;140(2):215-20. doi: 10.1016/j.ygyno.2015.12.007. Epub 2015 Dec 12. PMID 26691222
- [Background] Lim MC, Lee HS, Jung DC, Choi JY, Seo SS, Park SY. Pathological diagnosis and cytoreduction of cardiophrenic lymph node and pleural metastasis in ovarian cancer patients using video-assisted thoracic surgery. Ann Surg Oncol. 2009 Jul;16(7):1990-6. doi: 10.1245/s10434-009-0486-5. Epub 2009 Apr 30. PMID 19408045
- [Background] Yoo HJ, Lim MC, Song YJ, Jung YS, Kim SH, Yoo CW, Park SY. Transabdominal cardiophrenic lymph node dissection (CPLND) via incised diaphragm replace conventional video-assisted thoracic surgery for cytoreductive surgery in advanced ovarian cancer. Gynecol Oncol. 2013 May;129(2):341-5. doi: 10.1016/j.ygyno.2012.12.023. Epub 2013 Jan 3. PMID 23290988
- [Derived] Park SJ, Na KJ, Lee M, Park IK, Chung HH, Kang CH, Kim JW, Park NH, Kim YT, Song YS, Park S, Kim HS. Impact of supradiaphragmatic lymphadenectomy on the survival of patients in stage IVB ovarian cancer with thoracic lymph node metastasis. Front Oncol. 2023 Aug 10;13:1203127. doi: 10.3389/fonc.2023.1203127. eCollection 2023. PMID 37637060